CLINICAL TRIAL: NCT02209441
Title: Phase I Study of Sorafinib With Folfox4 as First-line Treatment in Advanced/Metastatic Gastric Cancer
Status: Available | Type: Expanded Access
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Shi Yuankai, vice president, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Other Study IDs: BAY43
Record Dates: First submitted 2014-08-04; First posted 2014-08-06 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Gastric Cancer.
Keywords: sorafenib, gastric cancer, FOLFOX4
MeSH Terms: conditions — Stomach Neoplasms

INTERVENTIONS:
Drug: Phase I Dose-finding Study of Sorafenib Study

SUMMARY:
* To determine the maximum-tolerated dose (MTD) and dose-limiting toxicity (DLT) of sorafenib in combination with FOLFOX4 (oxaliplatin/leucovorin/5-fluorouracil) as first-line treatment for advanced gastric cancer
* The design of the study incorporated a standard 3 + 3 dose escalation procedure to guide elevation of the sorafenib dosage to the next level

DETAILED DESCRIPTION:
-Twice-daily dosing of sorafenib 200 mg in combination with FOLFOX4 proved effective and safe for the treatment of advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years.
* documented gastric adenocarcinoma via histological or cytological examinations;
* newly diagnosed or recurrent unresectable advanced and metastatic gastric cancer;
* no history of chemotherapy or radiation therapy; at least one lesion with a measurable diameter; -
* an Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1;
* an expected survival time of at least 3 months;
* and provision of informed consent by patients prior to commencement of the study.

Exclusion Criteria:

* a present or past medical history of other tumors, except for cured skin cancer (non-melanoma) or carcinoma in situ of the cervix;
* surgery, open biopsy, or obvious trauma within 28 days prior to enrolment; peritoneal seeding or intestinal obstruction;
* severe gastrointestinal bleeding; grade 1 or greater peripheral neuropathy
* a past medical history of serious neurological or psychiatric diseases; pregnancy or lactation;
* women of childbearing potential unwilling to use adequate contraception; a past medical history of heart disease such as greater than grade 2 New York Heart Association (NYHA) congestive heart failure, unstable coronary heart disease (patients having episodes of myocardial infarction earlier than 12 months prior to the study were allowed to enrol), arrhythmia requiring antiarrhythmic therapy (patients on β-blockers or digoxin were allowed to enrol), or uncontrolled hypertension; severe active infection
* epileptic patients requiring medical treatment (such as corticosteroids or antiepileptic drugs);
* patients who had received immunotherapy within 4 weeks prior to or throughout the study or had received mitomycin C or nitrourea drugs within 4 weeks previously;
* allergies or possible allergies to the study medications or other drugs administered during the study;
* any patient safety or compliance issues that might jeopardize their participation in the study;
* an inability to swallow oral drugs.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult